CLINICAL TRIAL: NCT02836730
Title: Long-term Outcomes of Surgical and Nonsurgical Management of Sciatica Secondary to a Lumbar Disc Herniation or Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: Back and Rehabilitation Center, Copenhagen (Other Government)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tom Petersen, Researcher, Back and Rehabilitation Center, Copenhagen
Other Study IDs: Kirurgi-1507-2016
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lumbar Disc Herniation; Lumbar Spinal Stenosis
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lumbar disc herniation: Patients with surgery for lumbar disc herniation;
  Interventions: Procedure: Low back pain surgery
- Spinal stenosis: Patients with surgery for lumbar spinal stenosis
  Interventions: Procedure: Low back pain surgery
- No surgery: Patients with no surgery for lumbar disc herniation; patients with no surgery for lumbar spinal stenosis;
  Interventions: Procedure: Low back pain surgery

INTERVENTIONS:
Procedure: Low back pain surgery

SUMMARY:
The rate of success 12 months after surgery is reported to be 60-65% in patients with lumbar disc herniation and 60-70% in patients with spinal stenosis.

At the Back Center Copenhagen, patients with persistent low back pain caused by lumbar disc herniation and spinal stenosis are treated by a multidisciplinary team comprising rheumatologists, physiotherapists, chiropractors, and social workers according to current guidelines. Therefore we have a unique opportunity to report the long term outcome in candidates for surgery, regardless of whether they have surgery or not, after having received optimal but unsuccessful nonsurgical treatment.

The purpose of this study is to answer the following questions: 1) What is the proportion of patients operated upon after referral to surgical evaluation with positive MRI findings, persistent low back pain, and poor outcome following non-operative treatment? 2) What was the outcome in these patients 2 years following referral? 3) Where any baseline variables predictive of good or poor postsurgical outcome? 4) Where there any difference in outcome in patients with or without surgery?

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms more than 3 months
* Positive imaging findings
* Non-surgical treatment unsuccessful

Exclusion Criteria:

* Age below 18 or above 65 years
* Lumbar fusion
* Psychiatric disorders
* Other serious diseases
* Unable to understand the Danish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain referred to surgical evaluation with positive MRI findings, persistent low back pain, and poor outcome following non-operative treatment
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2004-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Disability | 2 years follow-up
  Roland Morris Disability Questionnaire. lack of success is defined as less than 30% improvement

SECONDARY OUTCOMES:
Back og leg pain | 2 years follow-up
  10 point Numeric Rating Scales for current pain, worst pain and average pain. Lack of success defined as less than 30% improvement.
Global outcome | 2 years follow-up
  5 point Likert Scale. Lack of success is defined as a score of No change, Worse, or Much worse
Reoperation during follow-up | 2 years follow-up
  Self reporting by questionnare
Sick leave because of back pain | 2 years follow-up
  Self reporting by questionnare
Contacts to the health care system because of back pain | 2 years follow-up
  Self reporting by questionnare

CONTACTS AND LOCATIONS:
Locations (1):
- Back and Rehabilitation Center Copenhagen, Copenhagen, Copenhagen, Denmark